CLINICAL TRIAL: NCT02598076
Title: Motivational Interviewing to Enhance Adherence of Patients With Psychogenic Non-epileptic Seizures: A Model of Patient Engagement in Functional Neurological Symptom Disorders
Brief Title: Motivational Interviewing to Enhance Adherence of Patients With Psychogenic Non-epileptic Seizures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Academy of Neurology (Other)
Responsible Party: Principal Investigator, Benjamin Tolchin, Clinical Fellow, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001152
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Psychogenic Non-epileptic Seizures, Motivational Interviewing
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): Group will receive standard treatment for psychogenic non-epileptic seizures. They will undergo an initial clinic visit with a neuropsychiatrist and neurologists. They will not undergo any subsequent motivational interview. Following the initial clinic visit, all subjects with ongoing seizures will either be scheduled for ongoing psychotherapy for treatment of PNES at Brigham and Women's Hospital or referred to a local psychotherapist according to their preference.
  Interventions: Behavioral: standard psychotherapy
- MI (Experimental): Group will receive an initial clinic visit with a neuropsychiatrist and neurologists, identical to the initial clinic visit for the control group. In addition they will receive 1 session of motivational interviewing immediately following the initial clinic visit. These patients will be questioned using standardized motivational interviewing techniques by the study author who is a board certified neurologist and who has formal training and certification in motivational interviewing.
  Following the initial clinic visit, all subjects with ongoing seizures will either be scheduled for ongoing psychotherapy for treatment of PNES at Brigham and Women's Hospital or referred to a local psychotherapist according to their preference (identical treatment in control and MI arms).
  Interventions: Behavioral: motivational interviewing; Behavioral: standard psychotherapy

INTERVENTIONS:
Behavioral: motivational interviewing — Motivational interviews will include the classical 4 steps of MI: 1) engagement (in which the patient's goals and interests are elicited and the therapeutic alliance is established); 2) focusing (in which the specific subjects of discussion and intervention are negotiated); 3) strengthening motivation (in which the patients' reasons for healthcare intervention are made explicit, discussed, and reinforced); and 4) planning (in which actions for healthcare intervention are planned out based on the patients' own goals and interests). MI will be performed by the study author who is a board certified neurologist and who has formal training and certification in motivational interviewing.
  Arms: MI
Behavioral: standard psychotherapy — Standard cognitive behavioral therapy based psychotherapy for the treatment of PNES

SUMMARY:
All subjects will attend an initial clinic visit with the neuropsychiatrist and epileptologist. At the end of this visit, those subjects randomized to motivational interviewing will be questioned using standardized motivational interviewing techniques by the study author who is a board certified neurologist and who will have formal training and certification in motivational interviewing.

Those subjects randomized to the control group will also undergo an initial clinic visit with a neuropsychiatrist and neurologists. However they will not undergo any subsequent motivational interview. Following the initial clinic visit, all subjects with ongoing seizures will either be scheduled for ongoing psychotherapy for treatment of PNES at Brigham and Women's Hospital or referred to a local psychotherapist according to their preference.

All subjects will be contacted by phone at 3 month follow-up. If necessary they will be called 5 times at various times during the day and early evening. If they are not reached, they will receive a letter requesting them to contact the study staff to complete the study. Subjects will be questioned about their adherence to treatment. The primary outcome will be the number of psychotherapy sessions for the treatment of PNES in which they have participated over the past three months. They will also be assessed for secondary outcomes including dichotomous adherence (either seizure freedom or active participation in psychotherapy for the treatment of PNES, with more than 5 sessions over the past 3 months), seizure frequency over the past month, number of hospitalizations and emergency department visits over the past 3 months, and quality of life as measured by the brief QOLIE-10 instrument. For those patients who give permission, their psychotherapists will be contacted by study staff to confirm the exact number of psychotherapy sessions over the past 3 months. A standard Partners clinical records release form with the patient's signature will be sent to the therapist's office.

DETAILED DESCRIPTION:
Specific Aim: To determine whether motivational interviewing improves adherence to treatment (primary outcome), seizure frequency, healthcare usage, and quality of life (secondary outcomes).

Hypothesis: A brief in-person interview, using motivational interviewing techniques in addition to standard psychotherapy, will improve adherence, seizure frequency, healthcare usage, and quality of life at 6-month follow-up among patients with PNES when compared to a control group receiving only standard psychotherapy.

Baseline demographic data, psychiatric comorbidities, seizure frequency, quality of life, and healthcare resource utilization will be recorded following enrollment during the inpatient stay as part of PHRC IRB protocol 2013P000133. If the patient is not enrolled in protocol 2013P000133, baseline demographic data, seizure data, psychiatric comorbidities, qualities of life and healthcare resource utilization will be collected during the admission at which the patient is diagnosed. All enrolled subjects will be scheduled for an initial appointment in the joint psychiatry-neurology clinic with a board certified neuropsychiatrist and board certified neurologists, which is standard of care for newly diagnosed PNES patients at Brigham and Women's Hospital.

All subjects will attend the initial clinic visit with the neuropsychiatrist and epileptologist. At the end of this visit, those subjects randomized to motivational interviewing will be questioned using standardized motivational interviewing techniques by the study author who is a board certified neurologist and who will have formal training and certification in motivational interviewing.

Motivational interviews will include the classical 4 steps of MI:

1. engagement (in which the patient's goals and interests are elicited and the therapeutic alliance is established);
2. focusing (in which the specific subjects of discussion and intervention are negotiated);
3. strengthening motivation (in which the patients' reasons for healthcare intervention are made explicit, discussed, and reinforced); and
4. planning (in which actions for healthcare intervention are planned out based on the patients' own goals and interests).

The initial clinic visit and subsequent interview will be recorded with the patients' consent, and blinded reviewers hired through the department of psychiatry, trained and certified in motivational interviewing, will score the audio recordings using the Motivational Interviewing Treatment Integrity code (MITI) 4.0 to assess fidelity to standardized motivational interviewing techniques. Recordings and blinded review of interviews are for the sole purpose of ensuring that the interviewer is in fact using proper interviewing techniques (ie motivational interviewing techniques for patients in the motivational interviewing arm and abstinence from motivational interviewing techniques in the control arm). Such recordings and review are recommended in motivational interviewing research.

Those subjects randomized to the control group will also undergo an initial clinic visit with a neuropsychiatrist and neurologists - again recorded with the subjects' consent and scored using the MITI 4.0 to assess abstinence from motivational interviewing techniques. However they will not undergo any subsequent motivational interview. Following the initial clinic visit, all subjects with ongoing seizures will either be scheduled for ongoing psychotherapy for treatment of PNES at Brigham and Women's Hospital or referred to a local psychotherapist according to their preference.

All subjects will be contacted by phone at 3 month follow-up. If necessary they will be called 5 times at various times during the day and early evening. If they are not reached, they will receive a letter requesting them to contact the study staff to complete the study. Subjects will be questioned about their adherence to treatment. The primary outcome will be the number of psychotherapy sessions for the treatment of PNES in which they have participated over the past three months. They will also be assessed for secondary outcomes including dichotomous adherence (either seizure freedom or active participation in psychotherapy for the treatment of PNES, with more than 5 sessions over the past 3 months), seizure frequency over the past month, number of hospitalizations and emergency department visits over the past 3 months, and quality of life as measured by the brief QOLIE-10 instrument. For those patients who give permission, their psychotherapists will be contacted by study staff to confirm the exact number of psychotherapy sessions over the past 3 months. A standard Partners clinical records release form with the patient's signature will be sent to the therapist's office.

ELIGIBILITY:
Inclusion Criteria:

* The study population will be screened from all patients diagnosed with PNES in Brigham and Women's Hospital by capture of a definitive event on video EEG without EEG correlate.
* Patients with a mixed diagnosis of both PNES and epileptic seizures will be included.

Exclusion Criteria:

* Pediatric patients (under age 18) are not evaluated by EEG in our hospital and will therefore be excluded
* Estimated IQ<70
* Active substance use disorder
* Pregnancy or active medical issues anticipated to preclude participation in weekly psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Dworetzky, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Interviewing: Group will receive an initial clinic visit with a neuropsychiatrist and neurologists, identical to the initial clinic visit for the control group. In addition they will receive 1 session of motivational interviewing immediately following the initial clinic visit. These patients will be questioned using standardized motivational interviewing techniques by a board certified neurologist with formal training and certification in motivational interviewing.
  Following the initial clinic visit, all subjects with ongoing seizures will either be scheduled for ongoing psychotherapy for treatment of PNES at BWH or referred to a local psychotherapist according to their preference.
  motivational interviewing: Motivational interviews will include the classical 4 steps of MI: 1) engagement; 2) focusing; 3) strengthening motivation; and 4) planning.
  standard psychotherapy: Standard cognitive behavioral therapy based psychotherapy for the treatment of PNES
Period: Overall Study
Arm/Group | Control | Motivational Interviewing
Started | 31 | 29
Completed | 29 | 26
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Motivational Interviewing | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (14.3) | 39.6 (16.8) | 40.2 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 3 | 3 | 6
  Hispanic | 7 | 6 | 13
  White, non-Hispanic | 20 | 20 | 40
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
years of education [Mean (Standard Deviation); unit: years] — Population: participant unwilling to complete baseline questionnaire
  years
    number analyzed (Participants) | 31 | 28 | 59
    (all) | 13.8 (2.5) | 13.0 (2.7) | 13.4 (2.6)
household income [Median (Inter-Quartile Range); unit: dollars] — Population: participants unwilling to provide information
  dollars
    number analyzed (Participants) | 19 | 21 | 40
    (all) | 42000 [19200 to 100000] | 30000 [16000 to 70000] | 33000 [17375 to 95000]
major depressive disorder [Count of Participants; unit: Participants] — Population: participant unwilling to provide information
  Participants
    number analyzed (Participants) | 31 | 28 | 59
    (all) | 13 | 12 | 25
generalized anxiety disorder [Count of Participants; unit: Participants] — Population: participant unwilling to complete baseline questionnaire
  Participants
    number analyzed (Participants) | 31 | 28 | 59
    (all) | 19 | 15 | 34
Post traumatic stress disorder [Count of Participants; unit: Participants] — Population: participant unwilling to provide information
  Participants
    number analyzed (Participants) | 31 | 28 | 59
    (all) | 10 | 12 | 22
History of abuse [Count of Participants; unit: Participants] — Population: participant unwilling to provide information
  Participants
    physical abuse: number analyzed (Participants) | 31 | 28 | 59
    physical abuse | 11 | 11 | 22
    sexual abuse: number analyzed (Participants) | 31 | 28 | 59
    sexual abuse | 15 | 13 | 28
    emotional abuse: number analyzed (Participants) | 31 | 28 | 59
    emotional abuse | 11 | 11 | 22
    any abuse: number analyzed (Participants) | 31 | 28 | 59
    any abuse | 18 | 18 | 36
delay to diagnosis of PNES [Median (Inter-Quartile Range); unit: months] — Population: participant unwilling to provide information
  months
    number analyzed (Participants) | 31 | 28 | 59
    (all) | 3 [1 to 37] | 9 [2 to 57] | 7 [1 to 48]
psychogenic seizure frequency [Median (Inter-Quartile Range); unit: PNES per week] — participant unwilling to provide information Population: participant unwilling to provide information
  PNES per week
    number analyzed (Participants) | 31 | 28 | 59
    (all) | 3 [1 to 7] | 4 [1 to 16] | 4 [1 to 8]
Quality of Life in Epilepsy (QOLIE)-10 [Mean (Standard Deviation); unit: units on a scale] — Quality of Life in Epilepsy (QOLIE)-10 scale is a validated, reliable instrument measuring quality of life on a scale from 10 (best) to 50 (worst). Total score was used. No sub-scales were used. Population: participants unwilling to complete instrument
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 28.0 (9.5) | 28.4 (8.8) | 28.2 (9.0)
Emergency Department visits per month [Median (Inter-Quartile Range); unit: visits per month] — Population: participants unwilling to provide information
  visits per month
    number analyzed (Participants) | 28 | 26 | 54
    (all) | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]
referred to psychotherapy at Brigham and Women's Hospital [Count of Participants; unit: Participants] | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Patients are classified as adherent if they attend 8 or more of the recommended 12 weekly psychotherapy sessions over a 16 week period. Otherwise they are classified as non-adherent.
Time Frame: 4 months
Population: Analysis population includes all participants for whom follow-up data was available. Patients who were lost to contact (after 7 phone calls and a mailed letter) for whom follow-up data was not available, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Motivational Interviewing
Number analyzed (Participants) | 29 | 26
Participants | 9 | 17
Statistical Analysis 1: Comparison: Control vs Motivational Interviewing; Test type: Superiority; p = 0.015, t-test, 2 sided

2. Secondary Outcome: Percent Decrease in PNES Frequency
Description: Percent decrease in monthly PNES frequency
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline seizures
Arm/Group | Control | Motivational Interviewing
Number analyzed (Participants) | 28 | 26
percentage of baseline seizures | 34.8 (89.7) | 76.2 (39.2)
Statistical Analysis 1: Comparison: Control vs Motivational Interviewing; Test type: Superiority; p = 0.034, t-test, 2 sided

3. Secondary Outcome: Change in Number of Monthly Emergency Department Visits
Description: Change from baseline number of Emergency Department visits per month.
Time Frame: 4 months
Population: Participants who provided this data at 4 month telephone follow-up.
Measure: Mean (Standard Deviation); unit: ED visits per month
Arm/Group | Control | Motivational Interviewing
Number analyzed (Participants) | 28 | 26
ED visits per month | 0.06 (0.47) | -0.15 (0.76)
Statistical Analysis 1: Comparison: Control vs Motivational Interviewing; Test type: Superiority; p = 0.23, t-test, 2 sided

4. Secondary Outcome: PNES Freedom
Description: Patients are classified as PNES free if they have had no PNES in 3 months, otherwise they are classified as not PNES free.
Time Frame: 4 months
Population: Participants who provided information at 4 month telephone follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Motivational Interviewing
Number analyzed (Participants) | 28 | 26
Participants | 3 | 8
Statistical Analysis 1: Comparison: Control vs Motivational Interviewing; Test type: Superiority; p = 0.095, Fisher Exact

5. Secondary Outcome: Change in Quality of Life
Description: Change from baseline to 4 month follow-up, in quality of life in epilepsy (QOLIE)-10 score. Quality of Life in Epilepsy (QOLIE)-10 scale is a validated, reliable instrument measuring quality of life on a scale from 10 (best) to 50 (worst). Total score was used. No sub-scales were used.
Time Frame: 4 months
Population: Participants who provided QOLIE-10 information at 4-month follow-up
Measure: Mean (Standard Deviation); unit: units on QOLIE-10 scale
Arm/Group | Control | Motivational Interviewing
Number analyzed (Participants) | 23 | 24
units on QOLIE-10 scale | 1.8 (7.9) | 7.2 (10.0)
Statistical Analysis 1: Comparison: Control vs Motivational Interviewing; Test type: Superiority; p = 0.047, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Control | Motivational Interviewing
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT02598076/Prot_SAP_000.pdf